CLINICAL TRIAL: NCT00067639
Title: Pegfilgrastim (Neulasta) for Mobilization of Peripheral Blood Progenitor Cells (PBPC) in Patients With Multiple Myeloma
Brief Title: Pegfilgrastim (Neulasta) for Stem Cell Mobilization in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ID03-0164
Record Dates: First submitted 2003-08-25; First posted 2003-08-26 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; PBSC mobilization; Pegfilgrastim; Neulasta; PEG-G-CSF
MeSH Terms: conditions — Multiple Myeloma | interventions — pegfilgrastim; pegylated granulocyte colony-stimulating factor, human; Blood Component Removal; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegfilgrastim + Apheresis (Experimental): 12 mg Pegfilgrastim as subcutaneous injection on day 1 + Apheresis daily till target stem cell dose reached.
  Interventions: Drug: Pegfilgrastim (Neulasta); Procedure: Apheresis

INTERVENTIONS:
Drug: Pegfilgrastim (Neulasta) — 12 mg single injection of pegfilgrastim under the skin prior to apheresis.
  Other Names: PEG-G-CSF
Procedure: Apheresis — Collection of stem cells, repeated daily until target stem cell dose reached, maximum of 5 procedures.
  Other Names: Leukapheresis

SUMMARY:
In recent years PBPC have replaced bone marrow as the source of hematopoietic stem cells for autologous transplantation. One of the cited advantages of this procedure is the avoidance of bone marrow harvest, which frequently requires general anesthesia. Other advantages include faster neutrophil and platelet engraftment times, faster immune recovery, decrease in the amount of tumor contamination and technical ability to obtain stem cells from patients previously considered unharvestable because of marrow fibrosis or because of prior radiotherapy to the pelvis. Filgrastim has emerged as the preferred cytokine for stem cell mobilization based on its safety profile and the positive experience in granulocyte donors however, the number of circulating CD34+ cells does not occur until the third day after starting filgrastim injections. Pegfilgrastim stimulates the production and maturation of neutrophil precursors and enhances the functions of mature neutrophils in the same manner as filgrastim. Data form normal volunteers and in studies of patients with cancer have shown prolonged serum levels of the cytokine, with "self-regulation" of pegfilgrastim levels as a function of the neutrophil count. This confers a therapeutic advantage in clinical settings by allowing a less frequent dosing.

DETAILED DESCRIPTION:
Stem cells are a special type of blood cell, which are able to grow and divide. Stem cells are given to patients after high dose chemotherapy to help restore blood production and immunity. For an autologous stem cell transplant, stem cells are collected from a patient before they have chemotherapy, then they are "transplanted" back to the same patient after treatment. Circulating blood contains a very small number of stem cells. It is often necessary to use the drug NeupogenTM, by injection under the skin twice a day for three days, before stem cells are collected to help move the stem cells out of the bone marrow and into the circulating blood. When the stem cells are in the blood, they can be collected more easily. The study drug pegfilgrastim is very similar to NeupogenTM, however, it is longer lasting. Therefore, treatment can be given as a single injection rather than several injections over many days.

For this study, you will receive a single injection of pegfilgrastim under the skin. Starting 3 days after the injection, you will have blood tests (1-2 tablespoons) once a day. These blood tests will be used to learn if there are enough stem cells circulating in the blood to start the collection procedure and for tests to check for any side effects of the drug. These once a day blood tests will continue up to 10 days after the completion of the stem cell collection procedure. When the stem cell count reaches a certain level (usually 4 or 5 days after the injection), stem cell collection will be started and done once a day until enough cells have been collected for transplantation.

Before the collection starts, you will have blood (1-2 tablespoons) and urine samples collected for routine tests. You will also have a chest x-ray and an electrocardiogram (ECG - a test that measures the electrical activity of the heart). These tests are being done to make sure you can handle the collection process. You will then have a central venous line (CVL) placed. For this procedure, you will have a catheter (small flexible tube) placed in a large vein under the collar bone. The CVL will be used to collect the stem cells.

You will have your stem cells collected by a procedure called apheresis. This procedure is similar to donating platelets in a blood bank. In this process blood is collected through the CVL and is passed through a cell separator machine. White cells (that contain the stem cells) are collected and frozen and the remaining blood is given back to you. During the apheresis procedure blood is kept from clotting by a continuous injection of ACD-A (sodium citrate solution). This may cause some loss of calcium from the blood. To help with this side effect, a calcium containing solution is continuously injected during the process of stem cell collection. The procedure takes around 4-6 hours. If sufficient numbers of stem cells are not collected in a single procedure, the procedure is repeated until the required number of stem cells can be collected. The maximum number of procedures will be 5. If enough stem cells cannot be collected after 5 procedures you will be taken off the study and your doctor will discuss other treatment options with you.

The stem cells that are collected will be "transplanted" back to you after you have high-dose chemotherapy as part of your standard care.

This is an investigational study. Pegfilgrastim is FDA approved and is commercially available. It is approved to increase white blood cell count after chemotherapy. However, its use in the collection of stem cells for transplantation is experimental. Up to 48 participants will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Age 18 years or older
2. Patients with multiple myeloma undergoing autologous peripheral blood stem cell transplantation and PBPC cell collection without chemopriming.
3. Zubrod performance status < 3 (Appendix E)
4. Serum bilirubin < 1.5 times the upper limit of normal, serum SGOT and SGPT < 2 times the upper limit of normal, serum creatinine < 2.0 mg/dl
5. WBC > 3,500/ul
6. Platelet count > 100,000/ul prior to first apheresis procedure
7. Patients should not have received prior chemotherapy. Only patients who have been treated with thalidomide, bortezomib, +/- dexamethasone will be eligible.
8. Sufficient peripheral venous access or central venous catheter
9. Informed consent

Exclusion Criteria:

1. Serious intercurrent medical illness
2. History of bleeding disorders (except patients with treated, myeloma related bleeding disorders)
3. Untreated hypercoagulation abnormalities
4. Patients with prior history of pulmonary embolism, deep venous thrombosis requiring anticoagulant therapy, or placement of a venous filter.
5. Untreated symptomatic cardiac disease defined as left ventricular EF of <40% and NYHA functional class of > II (Appendix F)
6. Uncontrolled infection defined as fever or antibiotics within 72 hours of registration.
7. History of allergy to filgrastim, pegfilgrastim or known hypersensitivity to E-coli derived proteins.
8. Palpable splenomegaly or craniocaudal spleen length greater than 12 cms
9. Pregnancy
10. Use of aspirin, ibuprofen containing products within 7 days of enrollment
11. History of uncontrolled autoimmune disorder
12. Sickle cell trait/sickle cell disease
13. Women who are lactating or breast feeding
14. 14. Patients with abnormal cytogenetics that may be secondary to myelodysplasia (-5, -7 and 11q23 abnormalities) will be excluded
15. Peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of pegfilgrastim in mobilizing progenitor cells | Baseline to 10 days after pegfilgrastim injection

CONTACTS AND LOCATIONS:
Overall Officials: Chitra Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org